CLINICAL TRIAL: NCT05667649
Title: Ph 1, Open-Label Safety Study of Escalating Doses of Intracerebroventricular Injections of Ex Vivo Expanded, Autologous ADSCs in Participants With Mild-Moderate AD Whose Treatment is Not Addressed Adequately by Available Therapy
Brief Title: Autologous Activated Adipose-derived Stem Cells (RB-ADSC) Injected Directly Into the Brain for Mild to Moderate Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneration Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RB-ADSC-02
Record Dates: First submitted 2022-12-01; First posted 2022-12-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; AD; Autologous; Stem cells
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- RB-ADSC low dose (Experimental): Participants will receive one dose of 2x10^6 RB-ADSC infused in the previously implanted Ommaya reservoir
  Interventions: Biological: RB-ADSC
- RB-ADSC medium dose (Experimental): Participants will receive one dose of 5x10^6 RB-ADSC infused in the previously implanted Ommaya reservoir
  Interventions: Biological: RB-ADSC
- RB-ADSC high dose (Experimental): Participants will receive one dose of 10x10^6 RB-ADSC infused in the previously implanted Ommaya reservoir
  Interventions: Biological: RB-ADSC

INTERVENTIONS:
Biological: RB-ADSC — Ex Vivo Expanded, Autologous Adipose-Derived Stem Cells (ADSCs)

SUMMARY:
This is a research study to evaluate the safety of an investigational autologous cell product obtained from participant's own adipose tissue as a possible treatment for Alzheimer disease.

DETAILED DESCRIPTION:
This is a Phase 1, Open-Label Safety Study of Escalating Doses of Intracerebroventricular Injections of Ex Vivo Expanded, Autologous Adipose-Derived Stem Cells (ADSCs) in Participants with Mild to Moderate Alzheimer's Disease (AD) whose Treatment is not Addressed Adequately by Available Therapy (i.e., an unmet medical need). The investigational product, which is referred to as RB-ADSC, consists of stem cells obtained from the participant's own adipose tissue by lipoaspirate. After collection, the stem cells are cultured and expanded outside the body, and then reintroduced into the same patient. A soft plastic reservoir (Ommaya reservoir) is implanted under the scalp, communicating with the brain cavities (ventricles). This study will primarily evaluate the safety of RB-ADSC injected in the Ommaya reservoir in a 3 + 3 dose escalation study. The planned enrollment will be 9 participants, 3 participants per escalation Cohort.

The primary objectives will evaluate adverse events, serious adverse events, and dose limiting toxicities to determine a recommended phase 2 clinical trial dose. Secondary objectives will evaluate preliminary efficacy measured by clinical assessments, volumetric MRI (Neuro Quant®), CSF biomarkers (Phospho-Tau, Total Tau, AB-42), and diagnostic imaging comparison (Amyloid PET). Each participant will be followed for 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥45 and ≤80 years of age
* Mild to moderate AD diagnosis
* Adequate cognitive function
* Non-remarkable clinical laboratory
* Ability to voluntarily provide written informed consent
* No tumors or other disease responsible for dementia
* Well-controlled comorbidities, on stable medications for 3 months
* The participant is otherwise in good general health
* The participant must have a relative/caregiver
* Participant must be able to donate adequate amount of lipoaspirate to establish the final product
* Caregiver separately meets the specified inclusion/exclusion criteria for caregivers

Exclusion Criteria:

* Taking other medications for AD, except that donepezil memantine, AChEIs including patches, Vitamin E, fish oil, and/or gingko biloba are allowed if doses have been stable for at least 3 months prior to the Screening visit
* Stem cell implantation of any type within 3 months
* Existing ventriculoperitoneal shunts
* Neurological disorders except AD
* Psychiatric disorders including schizophrenia, bipolar/unipolar depressive disorder, delirium
* Drug or alcohol abuse or dependence within the past 5 years
* Participants with a history of cancer in the past 5 years
* No caregiver available to meet the inclusion criteria for caregivers

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The safety of RB-ADSC treatment in study participants with AD | up to 28 weeks
  Safety will be determined by incidence, type and severity of adverse events (AE) and serious adverse events (SAE) graded according to CTCAE v5.0 and CRS revised grading system and defined by clinical relevant findings at every visit and week 28 post-treatment in physical examination, vital signs and laboratory data

SECONDARY OUTCOMES:
Change from Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) | up to 52 weeks
  Measured by the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) is a cognitive performance test. The ADAS-cog score ranges from 0 to 70, with higher scores indicating greater cognitive impairment (higher score is worse outcome).
Change from Baseline in Mini Mental State Examination (MMSE) | up to 52 weeks
  Measured by the Mini Mental State Examination (MMSE). MMSE is a performance-based test of global cognitive status.. The MMSE score ranges from 0 to 30, with lower scores indicating greater cognitive impairment (lower score is worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duma C, Kopyov O, Kopyov A, Berman M, Lander E, Elam M, Arata M, Weiland D, Cannell R, Caraway C, Berman S, Scord K, Stemler L, Chung K, Khoudari S, McRory R, Duma C, Farmer S, Bravo A, Yassa C, Sanathara A, Singh E, Rapaport B. Human intracerebroventricular (ICV) injection of autologous, non-engineered, adipose-derived stromal vascular fraction (ADSVF) for neurodegenerative disorders: results of a 3-year phase 1 study of 113 injections in 31 patients. Mol Biol Rep. 2019 Oct;46(5):5257-5272. doi: 10.1007/s11033-019-04983-5. Epub 2019 Jul 20. PMID 31327120